CLINICAL TRIAL: NCT04851873
Title: A Phase IIIb, Open-label, Single-arm, Single-dose, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of Gene Replacement Therapy With Intravenous OAV101 (AVXS-101) in Pediatric Patients With Spinal Muscular Atrophy (SMA)
Brief Title: Safety and Efficacy of Intravenous OAV101 (AVXS-101) in Pediatric Patients With Spinal Muscular Atrophy (SMA)
Acronym: SMART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COAV101A12306; 2020-005995-37 (EudraCT Number)
Record Dates: First submitted 2021-04-06; First posted 2021-04-21 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Spinal Muscular Atrophy
Keywords: Zolgensma; OAV101; AVXS 101; gene therapy; Muscle atrophy; SBMA; spinal and bulbar muscular atrophy; spinal muscular atrophy; bulbar muscular atrophy; muscle function; myopathy; muscle wasting; atrophied muscle; loss of muscle strength
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Atrophy; Bulbo-Spinal Atrophy, X-Linked; Muscular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will receive a single administration of OAV101
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OAV101 (Experimental): Participants received a single IV dose administration of OAV101
  Interventions: Genetic: OAV101

INTERVENTIONS:
Genetic: OAV101 — Gene Therapy - 1.1e14 vector genome (vg)/kg as a one-time IV infusion was administered over approximately 60 minutes.

SUMMARY:
To evaluate the safety, tolerability and efficacy of intravenous administration of OAV101 (AVXS-101) in patients with spinal muscular atrophy (SMA) with bi-allelic mutations in the survival motor neuron 1 (SMN1) gene weighing ≥ 8.5 kg and ≤ 21 kg, over a 12 month period.

DETAILED DESCRIPTION:
This was an open-label, single arm, multi-center study designed to evaluate the safety, tolerability and efficacy of OAV101 in participants with SMA who weigh ≥ 8.5 kg and ≤ 21 kg. The study aimed to enroll approximately 24 to 30 participants, with approximately 6 to 10 participants across each of 3 weight brackets (8.5 to 13 kg, >13 to 17 kg, >17 to 21 kg).

Eligible participants received a single administration of OAV101 at the approved dose of 1.1e14 vg/kg on Day 1 (Treatment period), and were followed for a period of 12 months.

Participants were admitted to the hospital on Day -1 for pre-treatment baseline procedures. After receiving OAV101 on Day 1, participants underwent in-patient safety monitoring over the next 48 hours, after which the participant could be discharged, based on Investigator judgment.

After study completion, eligible participants could enroll into a Long Term follow-up study to collect additional safety and efficacy data. (COAV101A12308 (NCT05335876) https://classic.clinicaltrials.gov/ct2/show/NCT05335876?term=COAV101A12308&draw=2&rank=1))

ELIGIBILITY:
Inclusion

* Symptomatic SMA diagnosis based on gene mutation analysis with bi-allelic survival motor neuron 1 (SMN1) mutations (deletion or point mutations) and any copy of the survival motor neuron 2 (SMN2) gene.
* Weight ≥ 8.5 kg and ≤ 21 kg at the time of Screening Visit 2
* Naive to treatment or have discontinued an approved drug/therapy

Exclusion:

* Previous OAV101 use or previous use of any adeno-associated virus serotype 9 (AAV9) gene therapy
* BMI < 3rd percentile
* Participant with history of aspiration pneumonia or signs of aspiration
* Elevated anti-AAV9 antibody
* History of gene therapy, hematopoietic transplantation, or solid organ transplantation
* Inability to take corticosteroids
* Concomitant use of immunosuppressive therapy
* Requiring invasive ventilation, tracheostomy or awake non-invasive ventilation 9. Administration of vaccines 2 weeks prior to infusion of OAV101
* Awake hypoxemia or awake oxygen saturation level decrease
* Hepatic dysfunction
* Presence of a confirmed or suspected infection
* If previously treated with disease modifying therapy, specified washout times apply
* Documented any parental consanguinity.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (2):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
- Novartis Investigative Site, Randwick, New South Wales, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (2):
  - Novartis Investigative Site, Garches
  - Novartis Investigative Site, Strasbourg
- Novartis Investigative Site, Roma, RM, Italy
- Novartis Investigative Site, Lisbon, Portugal
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] McMillan HJ, Baranello G, Farrar MA, Zaidman CM, Moreno T, De Waele L, Jong YJ, Laugel V, Quijano-Roy S, Mercuri E, Chien YH, Straub V, Darras BT, Seibert J, Bernardo Escudero R, Alecu I, Freischlager F, Muntoni F; SMART Study Group. Safety and Efficacy of IV Onasemnogene Abeparvovec for Pediatric Patients With Spinal Muscular Atrophy: The Phase 3b SMART Study. Neurology. 2025 Jan 28;104(2):e210268. doi: 10.1212/WNL.0000000000210268. Epub 2024 Dec 30. PMID 39804575
- See also: If you have inquiries about possible participation in this clinical study, please go to this website, and select your region or country, to see if there is an investigator site near you. — https://medinfo.novartis.com/gene-therapies/
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 13 investigative sites across 9 countries.
Pre-assignment Details: The screening period began after signature of the study informed consent. The study included a screening period of up to 45 days. On Day -1, participants were admitted to the hospital for pre-treatment baseline procedures. On Day 1, participants received the study treatment.
Groups:
- OAV101 1.1e14 vg/kg 8.5-13 kg: 8.5-13 kg
- OAV101 1.1e14 vg/kg >13-17 kg: >13-17 kg
- OAV101 1.1e14 vg/kg >17-21 kg: >17-21 kg
Period: Overall Study
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg
Started | 7 | 8 | 9
Completed | 7 | 8 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg | Total
Number analyzed (Participants) | 7 | 8 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.027 (1.1458) | 4.519 (1.1769) | 6.137 (1.6018) | 4.690 (1.8240)
Age, Customized [Count of Participants; unit: Participants]
  0 < 28 days | 0 | 0 | 0 | 0
  28 days - < 2 years | 1 | 0 | 0 | 1
  2 years - < 12 years | 6 | 8 | 9 | 23
  12 years - <18 years | 0 | 0 | 0 | 0
  >= 18 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 4 | 3 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 1 | 6 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) by Weight Bracket
Description: An AE is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: Up to Month 12
Population: Safety set (The Safety Set comprised all participants who were administered investigational drug.)
Measure: Count of Participants; unit: Participants
Groups:
- OAV101 1.1e14 vg/kg Overall: Overall
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
Participants
  Any treatment-emergent adverse events | 7 | 8 | 9 | 24
  Any treatment-emergent adverse events related to OAV101 | 7 | 8 | 9 | 24
  Any severe treatment-emergent adverse events | 1 | 4 | 3 | 8
  Any serious treatment-emergent adverse events | 3 | 7 | 5 | 15
  Serious treatment-emergent adverse events related to OAV101 | 1 | 4 | 2 | 7
  Treatment-emergent adverse events leading to study discontinuation | 0 | 0 | 0 | 0
  Treatment-emergent adverse events leading to death | 0 | 0 | 0 | 0
  Treatment-emergent adverse events of special interest | 7 | 7 | 9 | 23

2. Primary Outcome: Number of Participants With Important Identified and Important Potential Risks (Adverse Events of Special Interest (AESI)) by Risk Name and Weight Bracket
Description: Important identified and important potential risks included the following AESIs: Hepatotoxicity, Thrombocytopenia, Cardiac adverse events, Dorsal root ganglia toxicity and Thrombotic microangiopathy.
  These were assessed by the investigator.
Time Frame: Up to Month 12
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
Participants
  Hepatotoxicity | 6 | 5 | 9 | 20
  Transient thrombocytopenia | 4 | 6 | 7 | 17
  Cardiac adverse events | 0 | 2 | 1 | 3
  Thrombotic microangiopathy | 0 | 0 | 0 | 0
  Dorsal root ganglia cell inflammation | 0 | 0 | 0 | 0

3. Primary Outcome: Summary of Participants Meeting Criteria for Potentially Clinically Significant Vital Sign Values by Weight Bracket - Systolic and Diastolic Blood Pressure
Description: Change from baseline in vital signs measurements - systolic and diastolic blood pressure (mmHg).
  Systolic Blood Pressure-Low:<=5th percentile of the age(Any Age), High:>=90th percentile of the age, gender, and height group (<18 yrs).
  Diastolic Blood Pressure-High:>=90th percentile of the age, gender, and height group(<18 yrs).
Time Frame: 12 months
Population: Safety set
Measure: Count of Participants; unit: Participants
Groups:
- OAV101 1.1e14 vg/kg >13-17kg: >13-17kg
- OAV101 1.1e14 vg/kg >17-21kg: >17-21kg
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
Participants
  Systolic Blood Pressure (mmHg) Low | 1 | 0 | 1 | 2
  Systolic Blood Pressure (mmHg) High | 7 | 8 | 8 | 23
  Diastolic Blood Pressure (mmHg) High | 7 | 7 | 8 | 22

4. Primary Outcome: Change From Baseline in Vital Signs Measurements - Systolic Blood Pressure (mmHg)
Time Frame: Baseline, Days 2 and 3, Weeks 1, 2, 3, 4, 6, 8, 10, 13, 26, 39 and 52
Population: Safety set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
mmHg
  Change from baseline at Day 2 | 5.3 (12.65) | -1.3 (13.01) | 0.4 (10.36) | 1.3 (11.75)
  Change from baseline at Day 3 | -2.3 (15.01) | -5.6 (11.16) | 3.0 (8.38) | -1.4 (11.62)
  Change from baseline at Week 1 | 13.4 (10.53) | -7.4 (15.59) | 2.0 (12.84) | 2.2 (15.18)
  Change from baseline at Week 2 | 11.7 (20.33) | -3.8 (17.60) | 1.8 (9.15) | 2.8 (16.45)
  Change from baseline at Week 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 3 (n=6,8,9,23) | 15.8 (8.04) | -3.5 (12.87) | -0.7 (7.25) | 2.7 (12.33)
  Change from baseline at Week 4 (n=6,8,8,22): number analyzed (Participants) | 6 | 8 | 8 | 22
  Change from baseline at Week 4 (n=6,8,8,22) | 12.3 (16.50) | -3.5 (15.89) | 6.8 (10.02) | 4.5 (15.05)
  Change from baseline at Week 6 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 6 (n=7,8,8,23) | 8.1 (12.92) | -2.8 (24.15) | 5.4 (15.39) | 3.4 (18.13)
  Change from baseline at Week 8 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 8 (n=7,7,9,23) | 3.9 (15.49) | -0.7 (14.57) | 3.6 (12.83) | 2.3 (13.69)
  Change from baseline at Week 10 | 10.0 (16.99) | -5.6 (13.19) | 4.6 (10.06) | 2.8 (14.32)
  Change from baseline at Week 13 | 6.1 (10.78) | -4.5 (17.50) | 1.4 (9.93) | 0.8 (13.28)
  Change from baseline at Week 26 | -5.7 (9.05) | -12.9 (15.34) | -6.9 (14.99) | -8.5 (13.46)
  Change from baseline at Week 39 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 39 (n=7,7,9,23) | 16.4 (29.70) | -10.3 (13.59) | -3.9 (3.56) | 0.3 (21.98)
  Change from baseline at Week 52 | 5.0 (21.60) | -7.8 (13.54) | 0.1 (10.81) | -1.1 (15.67)

5. Primary Outcome: Change From Baseline in Vital Signs Measurements - Diastolic Blood Pressure (mmHg)
Time Frame: Baseline, Days 2 and 3, Weeks 1, 2, 3, 4, 6, 8, 10, 13, 26, 39 and 52
Population: Safety set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
mmHg
  Change from baseline at Day 2 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Day 2 (n=6,8,9,23) | 1.7 (12.42) | 4.8 (13.22) | -2.1 (13.04) | 1.3 (12.71)
  Change from baseline at Day 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Day 3 (n=6,8,9,23) | -3.7 (12.29) | -5.1 (13.91) | 4.2 (5.45) | -1.1 (11.22)
  Change from baseline at Week 1 | 7.4 (20.07) | 1.8 (13.56) | 3.8 (13.41) | 4.2 (15.13)
  Change from baseline at Week 2 | 7.1 (16.07) | 7.3 (11.30) | 4.4 (10.33) | 6.2 (12.05)
  Change from baseline at Week 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 3 (n=6,8,9,23) | 12.0 (15.09) | -1.5 (14.01) | 5.0 (9.60) | 4.6 (13.28)
  Change from baseline at Week 4 (n=6,8,8,22): number analyzed (Participants) | 6 | 8 | 8 | 22
  Change from baseline at Week 4 (n=6,8,8,22) | 3.8 (19.27) | 1.8 (9.97) | 1.3 (8.53) | 2.1 (12.12)
  Change from baseline at Week 6 (n=6,8,8,22): number analyzed (Participants) | 6 | 8 | 8 | 22
  Change from baseline at Week 6 (n=6,8,8,22) | 10.3 (10.91) | -0.5 (17.87) | 6.5 (10.14) | 5.0 (13.77)
  Change from baseline at Week 8 (n=6,7,9,22): number analyzed (Participants) | 6 | 7 | 9 | 22
  Change from baseline at Week 8 (n=6,7,9,22) | 10.5 (14.57) | 3.0 (17.68) | 5.9 (11.72) | 6.2 (14.18)
  Change from baseline at Week 10 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 10 (n=6,8,9,23) | 6.7 (15.55) | -2.0 (8.88) | 4.8 (11.74) | 2.9 (12.01)
  Change from baseline at Week 13 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 13 (n=6,8,9,23) | 9.7 (15.37) | 0.4 (13.54) | 0.1 (11.03) | 2.7 (13.20)
  Change from baseline at Week 26 | -0.7 (9.05) | -9.1 (10.26) | -1.2 (7.55) | -3.7 (9.41)
  Change from baseline at Week 39 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 39 (n=7,7,9,23) | 2.4 (15.73) | -4.4 (13.01) | -0.4 (9.62) | -0.8 (12.44)
  Change from baseline at Week 52 | 0.3 (11.74) | -2.0 (11.89) | 1.7 (5.52) | 0.0 (9.60)

6. Primary Outcome: Change From Baseline in Vital Signs Measurements - Respiratory Rate (Breaths/Min)
Description: Change from baseline in vital signs measurements - Respiratory Rate (breaths/min)
Time Frame: Baseline, Days 2 and 3, Weeks 1, 2, 3, 4, 6, 8, 10, 13, 26, 39 and 52
Population: Safety set
Measure: Mean (Standard Deviation); unit: breaths/min)
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
breaths/min)
  Change from baseline at Day 2 | -1.1 (3.08) | -1.6 (3.74) | 0.8 (3.96) | -0.6 (3.66)
  Change from baseline at Day 3 | -0.1 (5.87) | -0.1 (4.52) | 0.4 (4.30) | 0.1 (4.66)
  Change from baseline at Week 1 | 2.7 (6.78) | -0.1 (4.22) | 1.6 (5.61) | 1.3 (5.45)
  Change from baseline at Week 2 | 2.4 (5.44) | -0.8 (5.01) | 1.4 (4.16) | 1.0 (4.81)
  Change from baseline at Week 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 3 (n=6,8,9,23) | 5.5 (8.96) | -1.8 (5.09) | 1.8 (5.02) | 1.5 (6.63)
  Change from baseline at Week 4 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 4 (n=7,8,8,23) | 2.6 (4.54) | 1.4 (7.35) | 1.4 (4.00) | 1.7 (5.31)
  Change from baseline at Week 6 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 6 (n=7,8,8,23) | 5.1 (9.56) | -0.6 (4.75) | 0.3 (6.43) | 1.4 (7.19)
  Change from baseline at Week 8 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 8 (n=7,7,9,23) | 3.3 (7.45) | -0.6 (4.47) | 0.0 (4.42) | 0.8 (5.52)
  Change from baseline at Week 10 | 3.3 (6.58) | -1.0 (4.31) | -0.3 (3.61) | 0.5 (4.99)
  Change from baseline at Week 13 | 1.7 (6.75) | -0.5 (3.51) | -0.6 (2.92) | 0.1 (4.44)
  Change from baseline at Week 26 | 4.1 (8.69) | 0.8 (3.69) | 0.7 (4.24) | 1.7 (5.71)
  Change from baseline at Week 39 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 39 (n=7,7,9,23) | 1.4 (5.03) | -1.7 (4.35) | -0.6 (4.56) | -0.3 (4.61)
  Change from baseline at Week 52 | 1.7 (7.34) | -0.5 (4.66) | -2.2 (3.19) | -0.5 (5.18)

7. Primary Outcome: Change From Baseline in Vital Signs Measurements - Pulse Rate (Beats/Min)
Description: Change from baseline in vital signs measurements - Pulse Rate (beats/min
Time Frame: Baseline, Days 2 and 3, Weeks 1, 2, 3, 4, 6, 8, 10, 13, 26, 39 and 52
Population: Safety set
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
beats/min
  Change from baseline at Day 2 | 3.3 (18.54) | 6.3 (4.43) | 16.3 (26.54) | 9.2 (19.35)
  Change from baseline at Day 3 | -1.4 (19.29) | -3.1 (14.21) | 10.2 (14.19) | 2.4 (16.36)
  Change from baseline at Week 1 | 1.4 (14.27) | -9.6 (18.04) | -3.9 (18.84) | -4.3 (17.19)
  Change from baseline at Week 2 | -13.4 (21.25) | -8.8 (15.21) | 4.7 (12.12) | -5.1 (17.39)
  Change from baseline at Week 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 3 (n=6,8,9,23) | 21.0 (21.83) | -3.8 (12.46) | 13.1 (15.12) | 9.3 (18.60)
  Change from baseline at Week 4 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 4 (n=7,8,8,23) | -4.7 (17.27) | -3.5 (22.82) | 12.8 (16.23) | 1.8 (19.95)
  Change from baseline at Week 6 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 6 (n=7,8,8,23) | 12.9 (20.70) | 0.0 (9.59) | 8.8 (17.64) | 7.0 (16.58)
  Change from baseline at Week 8 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 8 (n=7,7,9,23) | -3.6 (15.75) | -6.3 (22.69) | 6.4 (17.63) | -0.5 (18.83)
  Change from baseline at Week 10 | -3.9 (25.14) | -4.3 (16.57) | 9.7 (14.13) | 1.1 (19.08)
  Change from baseline at Week 13 | -6.4 (12.23) | 2.6 (15.65) | 8.4 (18.06) | 2.2 (16.28)
  Change from baseline at Week 26 | -6.9 (12.85) | -6.3 (17.00) | 3.8 (14.34) | -2.7 (15.12)
  Change from baseline at Week 39 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 39 (n=7,7,9,23) | -4.7 (21.85) | -7.7 (13.23) | 3.1 (17.12) | -2.6 (17.54)
  Change from baseline at Week 52 | -8.9 (10.32) | -16.4 (14.38) | 4.4 (16.46) | -6.4 (16.35)

8. Primary Outcome: Summary of Participants Meeting Criteria for Potentially Clinically Significant Vital Sign Values by Weight Bracket - Temperature
Description: Change from baseline in vital signs measurements - temperature (degrees Celsius)
  Temperature-Low:<=35ºC(Any Age),High:>=38.4ºC(<18 yrs).
Time Frame: 12 months
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
Participants
  Temperature (ºC) Low | 0 | 0 | 0 | 0
  Temperature (ºC) High | 1 | 0 | 1 | 2

9. Primary Outcome: Change From Baseline in Vital Signs Measurements - Temperature (Degrees Celsius)
Time Frame: Baseline, Days 2 and 3, Weeks 1, 2, 3, 4, 6, 8, 10, 13, 26, 39 and 52
Population: Safety set
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
degrees Celsius
  Change from baseline at Day 2 | 0.07 (0.502) | -0.11 (0.714) | 0.07 (0.918) | 0.01 (0.722)
  Change from baseline at Day 3 | 0.11 (0.261) | -0.48 (0.719) | 0.12 (0.319) | -0.08 (0.541)
  Change from baseline at Week 1 | -0.07 (0.386) | -0.44 (0.563) | 0.00 (0.548) | -0.17 (0.528)
  Change from baseline at Week 2 | 0.30 (0.592) | -0.41 (0.649) | -0.09 (0.478) | -0.08 (0.618)
  Change from baseline at Week 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 3 (n=6,8,9,23) | 0.32 (0.556) | -0.24 (0.403) | 0.02 (0.387) | 0.01 (0.474)
  Change from baseline at Week 4 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 4 (n=7,8,8,23) | 0.16 (0.673) | -0.31 (0.775) | 0.05 (0.431) | -0.04 (0.645)
  Change from baseline at Week 6 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 6 (n=7,8,8,23) | 0.26 (0.458) | -0.18 (0.599) | -0.09 (0.500) | -0.01 (0.535)
  Change from baseline at Week 8 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 8 (n=7,7,9,23) | 0.13 (0.547) | -0.21 (0.654) | 0.01 (0.386) | -0.02 (0.521)
  Change from baseline at Week 10 | 0.34 (0.351) | -0.45 (0.727) | 0.01 (0.553) | -0.05 (0.635)
  Change from baseline at Week 13 | 0.13 (0.399) | -0.06 (0.701) | 0.09 (0.473) | 0.05 (0.525)
  Change from baseline at Week 26 | 0.31 (0.453) | -0.15 (0.532) | 0.03 (0.324) | 0.05 (0.460)
  Change from baseline at Week 39 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 39 (n=7,7,9,23) | 0.33 (0.350) | -0.10 (0.622) | -0.11 (0.491) | 0.03 (0.518)
  Change from baseline at Week 52 | 0.63 (0.836) | -0.53 (0.819) | -0.11 (0.401) | -0.03 (0.814)

10. Primary Outcome: Change From Baseline in Vital Signs Measurements - Oxygen Saturation Level
Description: Change from baseline in vital signs measurements - oxygen saturation level (%).
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated+saturated) in the blood and then multiplied by 100.
Time Frame: Baseline, Days 2 and 3, Weeks 1, 2, 3, 4, 6, 8, 10, 13, 26, 39 and 52
Population: Safety set
Measure: Mean (Standard Deviation); unit: % Oxygen Saturated
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17kg | OAV101 1.1e14 vg/kg >17-21kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
% Oxygen Saturated
  Change from baseline at Day 2 | 0.0 (0.82) | -0.3 (1.04) | -0.4 (1.13) | -0.3 (0.99)
  Change from baseline at Day 3 | 0.3 (1.80) | -0.1 (0.83) | -1.3 (1.12) | -0.5 (1.41)
  Change from baseline at Week 1 | 0.1 (1.07) | -0.4 (2.00) | -0.8 (1.20) | -0.4 (1.47)
  Change from baseline at Week 2 | -0.7 (1.89) | -1.0 (1.51) | -0.8 (2.11) | -0.8 (1.79)
  Change from baseline at Week 3 (n=6,8,9,23): number analyzed (Participants) | 6 | 8 | 9 | 23
  Change from baseline at Week 3 (n=6,8,9,23) | -1.0 (1.90) | -0.3 (1.28) | -1.1 (1.05) | -0.8 (1.38)
  Change from baseline at Week 4 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 4 (n=7,8,8,23) | 0.0 (1.91) | -0.5 (1.31) | -0.8 (0.89) | -0.4 (1.38)
  Change from baseline at Week 6 (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Change from baseline at Week 6 (n=7,8,8,23) | -0.1 (1.21) | -1.0 (1.51) | -0.6 (1.19) | -0.6 (1.31)
  Change from baseline at Week 8 (n=7,7,9,23): number analyzed (Participants) | 7 | 7 | 9 | 23
  Change from baseline at Week 8 (n=7,7,9,23) | -0.7 (1.89) | 0.0 (1.15) | -0.4 (0.88) | -0.4 (1.31)
  Change from baseline at Week 10 | 0.3 (1.89) | -1.0 (1.93) | -0.7 (1.32) | -0.5 (1.72)
  Change from baseline at Week 13 | 0.1 (1.57) | -0.5 (1.07) | -0.4 (1.67) | -0.3 (1.43)
  Change from baseline at Week 26 | -0.6 (1.51) | -0.1 (1.36) | -0.2 (1.99) | -0.3 (1.60)
  Change from baseline at Week 39 (n=7,7,8,22): number analyzed (Participants) | 7 | 7 | 8 | 22
  Change from baseline at Week 39 (n=7,7,8,22) | -1.0 (1.41) | 0.1 (0.90) | -0.4 (1.19) | -0.4 (1.22)
  Change from baseline at Week 52 | -1.0 (2.00) | -0.6 (1.51) | -0.1 (1.54) | -0.5 (1.64)

11. Secondary Outcome: Achievement of Development Motor Milestones According to the Modified and Combined WHO-MGRS and Bayley Scale of Infant and Toddler Development.
Description: The World Health Organization-Multicentre Growth Reference Study (WHO-MGRS) and Bayley scale of Infant and Toddler Development was modified and combined into a single scale expressly for this study, to measure developmental motor milestones. These were assessed via the milestone checklist, formed of 10 yes/no questions with optional video documentation. The developmental milestones are: head control, sitting with support, sitting without support, sitting without support for 30 seconds, hands-and-knees crawling, pulls to stand, standing with assistance, walking with assistance, standing alone and walking alone. A yes response indicates that the patient reached a particular development milestone.
Time Frame: Baseline, Week 26 and Week 52
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 7 | 8 | 9 | 24
Participants
  Baseline Head control (Bayley GM #4) | 7 | 8 | 9 | 24
  Baseline Sits with support (Bayley GM #19) | 7 | 8 | 9 | 24
  Baseline Sitting without support (WHO MGRS) | 6 | 7 | 8 | 21
  Baseline Sits without support 30 s (Bayley GM #26) | 6 | 7 | 8 | 21
  Baseline Hands-and-knees crawling (WHO MGRS) | 1 | 3 | 6 | 10
  Baseline Pulls to stand (Bayley GM #35) | 1 | 3 | 5 | 9
  Baseline Standing with assistance (WHO MGRS) | 0 | 2 | 5 | 7
  Baseline Walking with assistance (WHO MGRS) | 0 | 2 | 5 | 7
  Baseline Standing alone (WHO MGRS) | 0 | 2 | 4 | 6
  Baseline Walking alone (WHO MGRS) | 0 | 2 | 4 | 6
  Week 26 Head control (Bayley GM #4) | 7 | 8 | 9 | 24
  Week 26 Sits with support (Bayley GM #19) | 7 | 8 | 9 | 24
  Week 26 Sitting without support (WHO MGRS) | 7 | 5 | 9 | 21
  Week 26 Sits without support 30 s (Bayley GM #26) | 7 | 5 | 8 | 20
  Week 26 Hands-and-knees crawling (WHO MGRS) | 2 | 3 | 6 | 11
  Week 26 Pulls to stand (Bayley GM #35) | 2 | 3 | 5 | 10
  Week 26 Standing with assistance (WHO MGRS) | 1 | 3 | 5 | 9
  Week 26 Walking with assistance (WHO MGRS) | 1 | 3 | 4 | 8
  Week 26 Standing alone (WHO MGRS) | 0 | 3 | 4 | 7
  Week 26 Walking alone (WHO MGRS) | 0 | 2 | 4 | 6
  Week 52 Head control (Bayley GM #4) | 7 | 8 | 9 | 24
  Week 52 Sits with support (Bayley GM #19) | 7 | 7 | 9 | 23
  Week 52 Sitting without support (WHO MGRS) | 7 | 7 | 8 | 22
  Week 52 Sits without support 30 s (Bayley GM #26) | 7 | 6 | 8 | 21
  Week 52 Hands-and-knees crawling (WHO MGRS) | 2 | 3 | 6 | 11
  Week 52 Pulls to stand (Bayley GM #35) (n=7,8,8,23): number analyzed (Participants) | 7 | 8 | 8 | 23
  Week 52 Pulls to stand (Bayley GM #35) (n=7,8,8,23) | 2 | 3 | 5 | 10
  Week 52 Standing with assistance (WHO MGRS) | 2 | 3 | 5 | 10
  Week 52 Walking with assistance (WHO MGRS) | 1 | 3 | 4 | 8
  Week 52 Standing alone (WHO MGRS) | 0 | 3 | 4 | 7
  Week 52 Walking alone (WHO MGRS) | 0 | 2 | 4 | 6

12. Secondary Outcome: Change From Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE), as Appropriate According to Participant Age
Description: The HFMSE was devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE is formed of 33 assessments. Each motor skill item is scored on a 3 point Likert scale from 0 (no response) to 2 (full response), with a total score range of 0 to 66. A higher score indicates a higher level of ability.
Time Frame: Baseline, Week 4, Week 13, Week 26, Week 39 and Week 52
Population: Participants in the Full Analysis Set (FAS) who had an available value for the outcome measure at the specified timepoints. The FAS includes all participants who were administered investigational drug.
Measure: Mean (Standard Deviation); unit: HFMSE total score on a scale
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg | OAV101 1.1e14 vg/kg Overall
Number analyzed (Participants) | 5 | 6 | 9 | 20
HFMSE total score on a scale
  Change from baseline at Week 4 (n=4,6,9,19): number analyzed (Participants) | 4 | 6 | 9 | 19
  Change from baseline at Week 4 (n=4,6,9,19) | 3.8 (2.99) | 2.3 (2.66) | 3.1 (3.10) | 3.0 (2.83)
  Change from baseline at Week 13 (n=4,6,9,19): number analyzed (Participants) | 4 | 6 | 9 | 19
  Change from baseline at Week 13 (n=4,6,9,19) | 1.3 (7.89) | 4.5 (3.99) | 3.9 (3.98) | 3.5 (4.83)
  Change from baseline at Week 26 (n=5,6,9,20) | 3.4 (5.18) | 4.3 (5.05) | 3.1 (4.14) | 3.6 (4.45)
  Change from baseline at Week 39 (n=5,5,9,19): number analyzed (Participants) | 5 | 5 | 9 | 19
  Change from baseline at Week 39 (n=5,5,9,19) | 2.6 (6.11) | -0.6 (4.72) | 4.3 (3.71) | 2.6 (4.87)
  Change from baseline at Week 52 (n=5,6,7,18): number analyzed (Participants) | 5 | 6 | 7 | 18
  Change from baseline at Week 52 (n=5,6,7,18) | 3.0 (5.24) | 3.7 (5.75) | 4.3 (4.07) | 3.7 (4.73)

13. Secondary Outcome: Change From Baseline in Revised Upper Limb Module (RULM), as Appropriate According to Participant Age.
Description: The RULM assesses motor performance in the upper limbs from childhood through adulthood in ambulatory and non-ambulatory individuals with SMA. 'The scale consists of an entry item to establish functional levels and 19 items covering distal to proximal movements. The entry item is a modified version of the Brooke scale, including activities ranging from no functional use of hands (score 0) to full bilateral shoulder abduction (score 6). The entry item does not contribute to the total score but serves as a functional classification of overall upper limb functional ability. Of the remaining 19 items, 18 are scored on a 3 point scoring system and 1 item is scored on a 2 point scoring system. The test is performed unilaterally using the limb preferred by the participant. The total score ranges from 0, if all the items cannot be performed, to 37, if all the activities are achieved fully without any compensation. ' Higher scores indicate higher levels of motor ability.
Time Frame: Baseline, Week 4, Week 13, Week 26, Week 39 and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: RULM total score on a scale
Groups:
- OAV101 1.1e14 vg/kg 8.5-13 kg Overall: Overall
Arm/Group | OAV101 1.1e14 vg/kg 8.5-13 kg | OAV101 1.1e14 vg/kg >13-17 kg | OAV101 1.1e14 vg/kg >17-21 kg | OAV101 1.1e14 vg/kg 8.5-13 kg Overall
Number analyzed (Participants) | 4 | 6 | 8 | 18
RULM total score on a scale
  Change from baseline at Week 4 | 2.8 (2.36) | 1.2 (1.33) | 1.0 (1.93) | 1.4 (1.89)
  Change from baseline at Week 13 | 4.3 (1.50) | 0.8 (2.32) | 2.0 (2.56) | 2.1 (2.52)
  Change from baseline at Week 26 | 5.3 (2.50) | 1.3 (1.21) | 1.6 (2.88) | 2.3 (2.74)
  Change from baseline at Week 39 (n=4,5,8,17): number analyzed (Participants) | 4 | 5 | 8 | 17
  Change from baseline at Week 39 (n=4,5,8,17) | 7.3 (2.22) | -0.6 (1.34) | 2.0 (4.34) | 2.5 (4.29)
  Change from baseline at Week 52 (n=3,6,8,17): number analyzed (Participants) | 3 | 6 | 8 | 17
  Change from baseline at Week 52 (n=3,6,8,17) | 6.0 (3.46) | 0.3 (1.63) | 1.8 (4.71) | 2.0 (4.02)

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the single dose of study treatment until end of study, up to maximum duration of 12 months
Groups:
- OAV101 1.1e14 vg/kg 8.5 to 13 kg: 8.5 to 13 kg
- OAV101 1.1e14 vg/kg Greater Than 13 to 17 kg: Greater than 13 to 17 kg
- OAV101 1.1e14 vg/kg Greater Than 17 to 21 kg: Greater than 17 to 21 kg
Arm/Group | OAV101 1.1e14 vg/kg 8.5 to 13 kg | OAV101 1.1e14 vg/kg Greater Than 13 to 17 kg | OAV101 1.1e14 vg/kg Greater Than 17 to 21 kg | OAV101 1.1e14 vg/kg Overall
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/9 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/7 | 7/8 | 5/9 | 15/24
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 9/9 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101 1.1e14 vg/kg 8.5 to 13 kg (N=7) | OAV101 1.1e14 vg/kg Greater Than 13 to 17 kg (N=8) | OAV101 1.1e14 vg/kg Greater Than 17 to 21 kg (N=9) | OAV101 1.1e14 vg/kg Overall (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Asthenia (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Subglottic laryngitis (Infections and infestations) | 1 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101 1.1e14 vg/kg 8.5 to 13 kg (N=7) | OAV101 1.1e14 vg/kg Greater Than 13 to 17 kg (N=8) | OAV101 1.1e14 vg/kg Greater Than 17 to 21 kg (N=9) | OAV101 1.1e14 vg/kg Overall (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 5
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Cushing's syndrome (Endocrine disorders) | 1 | 0 | 2 | 3
Cushingoid (Endocrine disorders) | 0 | 1 | 1 | 2
Blepharitis (Eye disorders) | 0 | 0 | 1 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0 | 1
Periorbital swelling (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 3 | 8
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 5 | 7 | 17
Malaise (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 5 | 10
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1 | 5 | 7
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 4 | 2 | 7
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 3
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1 | 5
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2 | 8
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Stoma site erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Torus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1
Blood potassium abnormal (Investigations) | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 0 | 2
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 1 | 2
Platelet count abnormal (Investigations) | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 3 | 2 | 2 | 7
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 3 | 2 | 1 | 6
Weight increased (Investigations) | 0 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 2 | 0 | 2
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 2 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT04851873/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT04851873/SAP_001.pdf